CLINICAL TRIAL: NCT05965258
Title: Improving Phenotypic Classification and Prediction of Treatment Outcomes in Patients With Non-ischemic Cardiomyopathy and Functional Mitral Regurgitation
Brief Title: Phenotypic Classification of FMR With CMR
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Deborah Kwon, MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 23-702; 1R01HL170090-01 (NIH)
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Nonischemic Congestive Cardiomyopathy; Functional Mitral Regurgitation; Ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Optimize mGDMT: NICM patients referred for mGDMT optimization
  Interventions: Diagnostic Test: Cardiac magnetic resonance (CMR)
- MitraClip and mGDMT: NICM patients who are fully medically optimized with significant FMR at the time of the baseline CMR and are referred for Mitraclip treatment
  Interventions: Diagnostic Test: Cardiac magnetic resonance (CMR)

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance (CMR) — Cardiac magnetic resonance (CMR) at 6 months. If referred to MitraClip, CMR will be performed at 6 months from the procedure.

SUMMARY:
The goal of the current research is to develop personalized risk prediction for functional mitral regurgitation (FMR) patients through explainable unsupervised phenomapping enriched with advanced cardiac magnetic resonance (CMR) imaging biomarkers, and to determine the CMR predictors of reverse remodeling following modern therapies for FMR.

The prospective study entails aiming to recruit 360 adult patients (ages >18 years) with EF 10-50% and FMR RF> 20%, who are clinically referred for CMR evaluation. Patients who enroll in our study will be referred for optimization of mGDMT and will undergo follow-up CMR studies at 6months. NICM patients who are fully medically optimized with significant FMR at the time of the baseline CMR and are referred for Mitraclip treatment will undergo follow-up CMR 6 months from Mitraclip intervention. NICM patients referred for mGDMT optimization, but have persistent or progressive FMR at the time of 6 month follow-up CMR and referred for Mitraclip therapy, will undergo a 2nd follow-up CMR 6 months from Mitraclip therapy.

DETAILED DESCRIPTION:
Functional mitral regurgitation (FMR) portends a bleak prognosis and is a common consequence of ischemic and non-ischemic cardiomyopathy (ICM, NICM), where adverse annular and left ventricular (LV) remodeling and/or infarction alters mitral valve (MV) function.

Prior studies demonstrate significant increases in mortality risk as severity of FMR increases; mortality rates range from 15-40% at 1 year. Furthermore, as the prevalence of heart failure (HF) is rising, FMR is projected to double from over 2 million patients in 2000 to over 4 million patients in the United States by 2030. Defining FMR severity, optimal timing of intervention, and most appropriate method for intervention remain controversial. Recently, MITRA-FR and COAPT trials demonstrated contrasting survival benefit with percutaneous MV repair, demonstrating the importance and need for more optimal selection criteria. Currently, the patient selection criteria for Mitraclip therapy are solely based on MV anatomy and controversial echocardiographic criteria for FMR severity. Cardiac magnetic resonance (CMR) provides an exciting opportunity to address numerous unmet needs regarding characterizing FMR and the need for more optimal selection criteria for improving outcomes. Superior accuracy and reproducibility for quantification of LV size and function, and gold standard tissue characterization, positions CMR as the ideal imaging modality for comprehensively characterizing FMR and the underlying myopathic processes that significantly impact response to FMR therapies. The goal of the current research is to develop personalized risk prediction for FMR patients through explainable unsupervised phenomapping enriched with advanced CMR imaging biomarkers, and to determine the CMR predictors of reverse remodeling following modern therapies for FMR.

The proposed research will leverage a large retrospective single center NICM CMR database. Our CMR NICM database currently features 458 NICM patients, who underwent CMR on a single CMR vendor platform from 2008-2017, who have been extensively curated with contoured data for standard CMR measures. An additional 802 NICM patients have been identified from our 2018-2021 CMR database with EF<50% with the same inclusion/exclusion criteria, which will be extensively curated to enable phenomapping discovery. An external 400 NICM patient cohort will be used as an external validation cohort.

The prospective study entails aiming to recruit 360 adult patients (ages >18 years) with EF 10-50% and FMR RF> 20%, who are clinically referred for CMR evaluation. Patients who enroll in our study will be referred for optimization of mGDMT with Heart Failure Pharmacist Clinic and followed every 2 weeks until optimized. All will return and undergo follow-up CMR studies at 6months. NICM patients who are fully medically optimized with significant FMR at the time of the baseline CMR and are referred for Mitraclip treatment will undergo follow-up CMR 6 months from Mitraclip intervention. NICM patients referred for mGDMT optimization, but have persistent or progressive FMR at the time of 6 month follow-up CMR and referred for Mitraclip therapy, will undergo a 2nd follow-up CMR 6 months from Mitraclip therapy. CMR will be done on dedicated cardiac research MRI scanner.

A ischemic cardiomyopathy subgroup will be assessed as a comparator cohort.

ELIGIBILITY:
Inclusion Criteria:

1 CMR LVEF <55% 2.FMR Fraction>20% or echo criteria consistent with at least moderate mitral regurgitation with adequate image quality

Exclusion Criteria:

1. >moderate aortic regurgitation/stenosis,
2. <18 years of age,
3. acute myocarditis,
4. eGFR<15
5. HCM
6. cardiac amyloidosis/sarcoidosis
7. prior mitral valve intervention
8. myocardial infarction within 8 weeks of CMR

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred to Cleveland Clinic Structural Interventional Cardiology Clinic for evaluation of possible percutaneous MV intervention are routinely referred for CMR as part of their clinical protocol, and will be recruited for this prospective study. Additionally, patients clinically referred for CMR for evaluation of cardiomyopathy, who are found to have FMR RF >20% for enrollment into this prospective study.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiac mortality, heart transplant, or LVAD implantation. | Up to 36 months
  Occurrence of cardiac mortality and/or heart transplant and/or LVAD implantation

SECONDARY OUTCOMES:
Change in FMR | 6 months
  a change of >5 units/percentage points compared to baseline
Change in NT-proBNP | 6 months
  30% change in NT-proBNP or decrease to level < 1000 compared to baseline
Change in KCQL score | 6 months
  5 point change in KCQL score compared to baseline
Change in 6-minute walk test | 6 months
  25 meter change in 6-minute walk test compared to baseline
Recurrent heart failure hospitalization | up to 1 year
  Occurrence of heart failure related hospitalization
Arrhythmias | up to 1 year
  Occurrence of arrhythmia
MI | up to 1 year
  Occurrence of myocardial infarction
Stroke | up to 1 year
  Occurrence of stroke
Heart transplant | up to 1 year
  Occurrence of heart transplant
LVAD implantation | up to 1 year
  Occurrence of implant of left ventricular assisted device (LVAD)
Mortality | up to 1 year
  Occurrence of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Kwon, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No